CLINICAL TRIAL: NCT04195802
Title: Self-administered Questionnaire to Evaluate Salt and Potassium Diet of Patients Followed in Nephrology - UniverSEL Study
Brief Title: Self-administered Questionnaire to Evaluate Salt and Potassium Diet of Patients Followed in Nephrology
Acronym: UniverSEL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL69_0458
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Nephropathy, Chronic Tubulointerstitial
MeSH Terms: conditions — Nephropathy, Chronic Tubulointerstitial | interventions — Salts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Salt and potassium Diet — Self-administration questionnary to evaluate the salt and potassium consumption

SUMMARY:
The aim of the study is to create a self-questionnaire to evaluate sodium and potassium diet in chronic kidney disease patients.

Questionnaires will be compared to 24h sodium and potassium urinary excretion (reference) A Bayesian network and a multiple regression will be used to select the most relevant items

ELIGIBILITY:
Inclusion Criteria:

* Adult consulting in nephrology and having a 24h sodium urinary excretion routinely determined
* Consent informed agreement

Exclusion Criteria:

* Do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult consulting in nephrology and having a 24h sodium urinary excretion routinely determined
Sampling Method: Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
The aim of the study is to create a self-administered questionnaire to evaluate sodium and potassium consumption in chronic kidney disease patients. | at inclusion
  comparison of answers to the self-questionnaire about salt and potassium diet with natriuresis and kaliuresis urinary excretion during 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre FAUVEL, MD, Principal Investigator — Service de néphrologie - HTA - Dialyse
Locations (1):
- Hôpital Edouard Herriot - Service de néphrologie - HTA - Dialyse, Lyon, France